CLINICAL TRIAL: NCT00385229
Title: Post Term Pregnancy - Induction of Labor or Monitoring of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REK 106-01
Record Dates: First submitted 2006-10-06; First posted 2006-10-09 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-11

CONDITIONS: Perinatal Morbidity
Keywords: Asphyxia neonatorum; Birth Injury; Meconium Aspiration Syndrome
MeSH Terms: conditions — Asphyxia Neonatorum; Birth Injuries; Meconium Aspiration Syndrome | interventions — Labor, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Induction (Experimental): induction of labor at gestational age 289(41 weeks+2 days)
  Interventions: Drug: induction of labor
- expectant management (No Intervention): expectant management at gestational age 289(41 weeks+2 days)

INTERVENTIONS:
Drug: induction of labor — Misoprostol, Dinoprostone, amniotomy, Oxytocin
  Arms: Induction

SUMMARY:
Post term pregnancy is a risk pregnancy. Aim of the study was to investigate whether induction of labor at gestational age 289(41 weeks+2 days) reduces neonatal morbidity compared to expectant management. Secondary aims was to assess the effect on mode of delivery and maternal complications, as well as assess women's views and experiences.

Our 0-hypothesis was that induction of labor at gestational age 41+2 did not result in better outcome of pregnancy, measured as perinatal morbidity.

Following inclusion, women were randomly allocated to induction of labor or to monitoring of pregnancy every third day until delivery

ELIGIBILITY:
Inclusion criteria:

* Routine ultrasound scan and delivery at St.Olav's Hospital
* Ability to speak Norwegian
* Singleton pregnancy
* Gestational age 289 +/- 2 days
* Cephalic presentation

Exclusion criteria:

- prelabor rupture of membranes

Sex: Female
Age Groups: Child, Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2002-09; Primary Completion 2003-12 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Neonatal morbidity | peri- en postnatal

SECONDARY OUTCOMES:
Maternal complications | peri- and postnatal
Mode of delivery | at birth
women's view | postpartum
Women's experiences | perinatal
Hormone levels | perinatal

CONTACTS AND LOCATIONS:
Overall Officials: Runa Heimstad, MD, Study Director — Department of Obstetrics, St.Olavs Hospital, Trondheim University Hospital
Locations (1):
- Department of Obstetrics, St.Olavs Hospital, Trondheim University Hospital, Trondheim, Norway

REFERENCES:
- [Result] Heimstad R, Skogvoll E, Mattsson LA, Johansen OJ, Eik-Nes SH, Salvesen KA. Induction of labor or serial antenatal fetal monitoring in postterm pregnancy: a randomized controlled trial. Obstet Gynecol. 2007 Mar;109(3):609-17. doi: 10.1097/01.AOG.0000255665.77009.94. PMID 17329511
- [Derived] Middleton P, Shepherd E, Morris J, Crowther CA, Gomersall JC. Induction of labour at or beyond 37 weeks' gestation. Cochrane Database Syst Rev. 2020 Jul 15;7(7):CD004945. doi: 10.1002/14651858.CD004945.pub5. PMID 32666584